CLINICAL TRIAL: NCT05356533
Title: Development of an Interactive, Web-based Drinking to Cope Intervention and Tools to Assess Coping Skill Utilization
Brief Title: Coping Skills for Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jennifer Cadigan, Assistant Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008998; 1R34AA028074 (NIH)
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Drinking; Coping Skills
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): A total of 60 young adults will be randomized to the 4-week, web-based drinking to cope intervention.
  Interventions: Behavioral: Drinking to Cope CBT skills
- Assessment Control (No Intervention): A total of 60 young adults will be randomized to the assessment only control condition.

INTERVENTIONS:
Behavioral: Drinking to Cope CBT skills — Young adults who drink to cope with negative affect will receive 8 web-based modules with cognitive behavioral skills
  Arms: Intervention

SUMMARY:
A total of 120 young adults who drink to cope with negative affect will be randomized to a 4-week, web-based intervention with interactive modules on cognitive-behavioral skills (n=60) or an assessment only control (n=60). Participants will complete 4 weekly assessments and a 1- and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

- Eligibility criteria at recruitment include: 1)18-25 years old; 2) Currently live in the state of WA, 3) Have a valid email address and phone number, 4) Drank alcohol at least once in the past month, 5) report at least 1 alcohol-related problem in the past month, 6) report using alcohol to cope with distress via negative reinforcement (i.e., to provide relief or reduction of stress or depressed mood) in the past month

Exclusion Criteria:

* None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Cadigan, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Assessment Control
Started | 60 | 60
Completed | 49 | 57
Not Completed | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Assessment Control | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.76 (2.095) | 21.84 (2.154) | 21.80 (2.117)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 50 | 53 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 13 | 22 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 36 | 22 | 58
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use-Peak Drinks
Description: Peak number of drinks; Item measuring peak alcohol consumption, "Think of the occasion you drank the most this past month. How much did you drink?", response options ranged from 0 (0 drinks) to 25 (25+ drinks);
Time Frame: past month
Measure: Mean (Standard Deviation); unit: number of drinks
Arm/Group | Intervention | Assessment Control
Number analyzed (Participants) | 48 | 56
number of drinks | 4.71 (3.25) | 4.79 (3.64)
Statistical Analysis 1: Comparison: Intervention vs Assessment Control; Test type: Superiority; p > .05, Mixed Models Analysis; Risk Ratio (RR) = 1.08
Statistical Analysis 2: Comparison: Intervention vs Assessment Control; Test type: Superiority; p > .05, ANOVA; Risk Ratio (RR) = 1.08

2. Primary Outcome: Alcohol Use-drinks Per Week
Description: The DDQ (Collins, Parks, & Marlatt, 1985) was used to measure the quantity of alcohol consumed by asking participants to estimate the typical number of drinks consumed on each day of the week, on average during the past month. A sum score of weekly total drinks per week was then calculated as the sum of the total number of drinks per week reported.
Time Frame: past month
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Intervention | Assessment Control
Number analyzed (Participants) | 48 | 56
drinks per week | 5.40 (5.51) | 6.09 (6.56)
Statistical Analysis 1: Comparison: Intervention vs Assessment Control; Test type: Superiority; p > .05, Mixed Models Analysis; Risk Ratio (RR) = 1.08

3. Primary Outcome: Alcohol Use-heavy Episodic Drinking
Description: Heavy Episodic Drinking; NIAAA item assessing binge drinking, "During the past month, how often did you have [4 or more drinks (for women) /5 or more drinks (for men)] containing any kind of alcohol within a two-hour period?", response options ranged from 0 (Never) to 7 (Every day);
Time Frame: past month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment Control
Number analyzed (Participants) | 49 | 57
score on a scale | 1.69 (0.92) | 1.79 (1.03)
Statistical Analysis 1: Comparison: Intervention vs Assessment Control; Test type: Superiority; p > .05, Mixed Models Analysis; Risk Ratio (RR) = 0.81

4. Primary Outcome: Alcohol Negative Consequences
Description: Alcohol Negative Consequences, Sum score (count) of negative consequences taken from Brief Young Adult Alcohol Consequences Questionnaire; Scores ranged from 0-24, with higher scores associated with more consequences.
Time Frame: Past Month
Measure: Mean (Standard Deviation); unit: number of consequences
Arm/Group | Intervention | Assessment Control
Number analyzed (Participants) | 48 | 55
number of consequences | 3.79 (4.70) | 4.64 (5.91)
Statistical Analysis 1: Comparison: Intervention vs Assessment Control; Test type: Superiority; p < .05, Mixed Models Analysis; Risk Ratio (RR) = 0.91

5. Primary Outcome: Alcohol Coping
Description: The Drinking Motives Questionnaire-Revised (DMQR; Grant V.V., Stewart S.H., O'Connor R.M., Backwell E., & Conrod P.J. (2007). Psychometric evaluation of the five-factor Modified Drinking Motives Questionnaire-Revised in undergraduates. Addictive Behaviors, 32(11), 2611-2632. Doi: 10.1016/j.addbeh.2007.07.004 ) was used to assess reasons for drinking. Using a 5-point scale (ranging from 'almost never/never' to 'almost always/always' participants rate how frequently they use alcohol for various reasons. The alcohol coping motives subscale was used which takes the average of the 9 items on the coping-depression subscale. Average scores ranged from 1-5, with higher scores are associated with greater use of coping.
Time Frame: Past Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment Control
Number analyzed (Participants) | 48 | 56
score on a scale | 1.24 (0.48) | 1.62 (0.86)
Statistical Analysis 1: Comparison: Intervention vs Assessment Control; Test type: Superiority; p > .05, Mixed Models Analysis; Risk Ratio (RR) = .99

6. Secondary Outcome: Depressive Symptoms
Description: depressive symptoms; The eight-item Patient Health Questionnaire depression scale (PHQ-8) was used to assess for symptoms of depression. A sum of the 8 items was used, with the summed score ranging from 0-24. Higher scores represent greater symptoms of depression.
Time Frame: Past month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment Control
Number analyzed (Participants) | 46 | 54
score on a scale | 6.98 (5.31) | 7.98 (5.41)
Statistical Analysis 1: Comparison: Intervention vs Assessment Control; Test type: Superiority; p > .05, Mixed Models Analysis; Risk Ratio (RR) = 1.11

ADVERSE EVENTS:
Time Frame: Data was collected over a 4 month period.
Description: The definition of adverse event and serious adverse event does not differ from the clinicialtrials.gov definition
Arm/Group | Intervention | Assessment Control
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT05356533/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT05356533/SAP_001.pdf